CLINICAL TRIAL: NCT03075787
Title: Cardiovascular Variability and Heart Rate Response Associated With Obstructive Sleep Apnea
Acronym: OSAS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1700176
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea; Heart rate; Heart rate variability; Microarousals; Autonomic nervous system activity
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with obstructive sleep apneas
  Interventions: Device: standard 24-h ambulatory polysomnography

INTERVENTIONS:
Device: standard 24-h ambulatory polysomnography — A standard 24-h ambulatory ad libitum polysomnography including EEG, electro-oculography (EOG), electromyography (EMG), EKG, was performed by a standard clinical.

SUMMARY:
Obstructive sleep apnea is often associated with microarousals and a stimulation of the sympathetic nervous system. The knowledge of this autonomic activation may help understanding the increase of cardiac risk observed in elderly. The aim of the study is to evaluate the relationship between obstructive sleep apnea severity, age, gender and heart rate response associated with obstructive sleep apnea. Drug-free patients diagnosed with obstructive sleep apneas were included. Clinical data and 24-h polysomnography recordings were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Restless legs syndrome patients
* Hospital routine for sleep disorders breathing diagnosis
* Apnea index > 0

Exclusion Criteria:

* Narcolepsy-cataplexy
* Sleep irregularities and sleep deprivation symptoms
* Lack of neurological or psychiatric diseases
* Periodic leg movements
* Central sleep apnea, treatment
* Cerebral lesion
* Medical illness
* Medication or drinks affecting sleep and wake state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive sleep apneas with a diagnosis from January 1st 2012 to September 1st 2016.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Amplitude of heart rate response associated with obstructive sleep apneas | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography

SECONDARY OUTCOMES:
Other Heart rate variability indices: Ptot | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography
Other Heart rate variability indices: very-low-frequency (VLF), low frequency (LF), low frequency normalized units (LFnu), high-frequency normalized units (HFnu) | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography
Other Heart rate variability indices: LF/HF | At diagnosis
  standard 24-h ambulatory ad libitum polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PICHOT, PhD, Study Chair — CHU SAINT-ETIENNE; Emilia SFORZA, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No